CLINICAL TRIAL: NCT04414449
Title: ICT-enabled Social-emotional Learning: Development of Responsibility and Well-being in the Educational Environment
Acronym: emoTIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Valencia (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, Inmaculada Montoya Castilla, Associate Professor, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PSI2017-84005-R
Record Dates: First submitted 2020-01-29; First posted 2020-06-04 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Adolescent - Emotional Problem
Keywords: Emotional Intelligence; Schools; Training Programs; Information and Communication Technologies (ICT)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): During the tutoring time, the intervention program is carried out in the experimental group, through emoTIC. EmoTIC is an emotional education program focused on the development of social-emotional competences through an application that can be used in mobile devices and tablets.
  Interventions: Other: ICT-enabled Social-emotional Learning
- Control group (No Intervention): During the period in which the intervention program is conducted in the experimental group, the control group will remain in the waitlist (will not participate in the intervention), and will carry out the program once the study is finished.

INTERVENTIONS:
Other: ICT-enabled Social-emotional Learning — ICT-enabled Social-emotional Learning
  Arms: Intervention group

SUMMARY:
The purpose of the study is to develop adolescents' social-emotional abilities to foster their personal and social responsibility, as well as their well-being, by means of a school-based intervention that addresses students, teachers and parents who participate in a social-emotional program using a technological platform. The program consists of activities based on solid theoretical frameworks on emotional intelligence, development of responsibility and meaningful learning.

DETAILED DESCRIPTION:
EmoTIC is an emotional education program focused on the development of social-emotional competences through an application that can be used in mobile devices and tablets.The program is based on a space adventure, and provides reinforcement through score points and more time for the additional games. The duration of the program is 8 weeks.

The emoTIC 8 version is designed so that teachers can easily carry it out in their classrooms. The application consists of application-guided activities that are put into practice in class, and includes other exercises that are meant to be carried out at home. The activities that are designed to be carried out during school hours are named "missions", and the exercises the students will do at home are called "trainings". Both are essential to adequately conduct the intervention.

The emoTIC SPACE version is designed so that it is carried out autonomously at home, through application-guided activities. This version includes 8 activities for each of the 4 areas.

ELIGIBILITY:
Inclusion Criteria:

* To have signed the informed consent (or their legal tutors).
* Being between 11 and 18 years old.

Exclusion Criteria:

* Inability to understand the activities or the language used.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Emotional Intelligence | Time 1 (first month)
  Trait Meta-Mood Scale (TMMS-24)
Emotional Intelligence | Time 2 (4th month)
  Trait Meta-Mood Scale (TMMS-24)
Emotional Intelligence | Time 3 (up to 1 year)
  Trait Meta-Mood Scale (TMMS-24)
Subjective Well-Being | Time 1 (first month)
  Life satisfaction and positive and negative affects
Subjective Well-Being | Time 2 (4th month)
  Life satisfaction and positive and negative affects
Subjective Well-Being | Time 3 (up to 1 year)
  Life satisfaction and positive and negative affects
Emotional Competence | Time 1 (first month)
  Emotional Skills and Competence Questionnaire
Emotional Competence | Time 2 (4th month)
  Emotional Skills and Competence Questionnaire
Emotional Competence | Time 3 (up to 1 year)
  Emotional Skills and Competence Questionnaire

SECONDARY OUTCOMES:
Somatic complaints | Time 1 (first month)
  The Somatic Complain List (SCL-10)
Somatic complaints | Time 2 (4th month)
  The Somatic Complain List (SCL-10)
Somatic complaints | Time 3 (up to 1 year)
  The Somatic Complain List (SCL-10)
Depression, Anxiety and Stress | Time 1 (first month)
  Depression, Anxiety and Stress Scale
Depression, Anxiety and Stress | Time 2 (4th month)
  Depression, Anxiety and Stress Scale
Depression, Anxiety and Stress | Time 3 (up to 1 year)
  Depression, Anxiety and Stress Scale
Psychosocial adjustment | Time 1 (first month)
  Strengths and Difficulties Questionnaire
Psychosocial adjustment | Time 2 (4th month)
  Strengths and Difficulties Questionnaire
Psychosocial adjustment | Time 3 (up to 1 year)
  Strengths and Difficulties Questionnaire
Suicide ideation | Time 1 (first month)
  "Sentia" Scale
Suicide ideation | Time 2 (4th month)
  "Sentia" Scale
Suicide ideation | Time 3 (up to 1 year)
  "Sentia" Scale
Personality | Time 1 (first month)
  Mini-Ipip Questionnaire
Personality | Time 2 (4th month)
  Mini-Ipip Questionnaire
Personality | Time 3 (up to 1 year)
  Mini-Ipip Questionnaire
Self-esteem | Time 1 (first month)
  Rosenberg Self-Esteem Scale
Self-esteem | Time 2 (4th month)
  Rosenberg Self-Esteem Scale
Self-esteem | Time 3 (up to 1 year)
  Rosenberg Self-Esteem Scale
Self-Efficacy | Time 1 (first month)
  General Self-Efficacy Scale
Self-Efficacy | Time 2 (4th month)
  General Self-Efficacy Scale
Self-Efficacy | Time 3 (up to 1 year)
  General Self-Efficacy Scale
School Social Climate | Time 1 (first month)
  Questionnaire to Assess School Social Climate (CECSCE)
School Social Climate | Time 2 (4th month)
  Questionnaire to Assess School Social Climate (CECSCE)
School Social Climate | Time 3 (up to 1 year)
  Questionnaire to Assess School Social Climate (CECSCE)
Social Responsibility | Time 1 (first month)
  Personal and Social Responsibility Questionnaire (PSRQ)
Social Responsibility | Time 2 (4th month)
  Personal and Social Responsibility Questionnaire (PSRQ)
Social Responsibility | Time 3 (up to 1 year)
  Personal and Social Responsibility Questionnaire (PSRQ)
Subjective Happiness | Time 1 (first month)
  Subjective Happiness Scale
Subjective Happiness | Time 2 (4th month)
  Subjective Happiness Scale
Subjective Happiness | Time 3 (up to 1 year)
  Subjective Happiness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Montoya-Castilla, PhD, Principal Investigator — Universitat de València
Locations (1):
- Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De la Barrera U, Postigo-Zegarra S, Monaco E, Gil-Gomez JA, Montoya-Castilla I. Serious game to promote socioemotional learning and mental health (emoTIC): a study protocol for randomised controlled trial. BMJ Open. 2021 Dec 31;11(12):e052491. doi: 10.1136/bmjopen-2021-052491. PMID 34972764
- [Derived] de la Barrera U, Monaco E, Postigo-Zegarra S, Gil-Gomez JA, Montoya-Castilla I. EmoTIC: Impact of a game-based social-emotional programme on adolescents. PLoS One. 2021 Apr 16;16(4):e0250384. doi: 10.1371/journal.pone.0250384. eCollection 2021. PMID 33861813